CLINICAL TRIAL: NCT01973634
Title: Comparison of Acute Toxicity and Cost Between Whole Breast Irradiation With Sequential Boost and Simultaneous Integrated Boost After Breast Conserving Surgery
Acronym: SeqB vs SIB
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2012/655
Record Dates: First submitted 2013-10-18; First posted 2013-10-31 (Estimated); Last update posted 2022-12-02 (Actual); Status verified 2022-11

CONDITIONS: Radiotherapy After Breast Conserving Surgery
Keywords: Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Minimal surgical margin 1 mm, conventional arm: seq boost (Active Comparator): Minimal surgical margin of 1 mm, conventional arm with sequential boost (15 x 2.67 Gy WBI + 4 x 2.5 Gy boost).
  Interventions: Radiation: sequential boost (15 x 2.67 Gy WBI + 4 x 2.5 Gy boost)
- Minimal surgical margin of 1 mm, experimental arm with SIB (Experimental): Minimal surgical margin of 1 mm, experimental arm with SIB (15 x 2.67 Gy WBI and SIB 15 x 2.67-3.12 Gy)
  Interventions: Radiation: SIB (15 x 2.67 Gy WBI and SIB 15 x 2.67-3.12 Gy)
- Minimal surgical margin <1 mm, conventional arm: seq boost (Active Comparator): Minimal surgical margin < 1 mm, conventional arm with sequential boost (15 x 2.67 Gy WBI + 6 x 2.48 Gy boost)
  Interventions: Radiation: sequential boost (15 x 2.67 Gy WBI + 6 x 2.48 Gy boost)
- Minimal surgical margin < 1 mm, experimental arm with SIB. (Experimental): Minimal surgical margin < 1 mm, experimental arm with SIB (15 x 2.67 Gy WBI and SIB 15 x 2.67-3.33 Gy)
  Interventions: Radiation: SIB (15 x 2.67 Gy WBI and SIB 15 x 2.67-3.33 Gy)

INTERVENTIONS:
Radiation: sequential boost (15 x 2.67 Gy WBI + 4 x 2.5 Gy boost) — Minimal surgical margin of 1 mm, conventional arm with sequential boost (15 x 2.67 Gy WBI + 4 x 2.5 Gy boost)
  Arms: Minimal surgical margin 1 mm, conventional arm: seq boost
Radiation: SIB (15 x 2.67 Gy WBI and SIB 15 x 2.67-3.12 Gy) — Minimal surgical margin of 1 mm, experimental arm with SIB (15 x 2.67 Gy WBI and SIB 15 x 2.67-3.12 Gy)
  Arms: Minimal surgical margin of 1 mm, experimental arm with SIB
Radiation: sequential boost (15 x 2.67 Gy WBI + 6 x 2.48 Gy boost) — Minimal surgical margin < 1 mm, conventional arm with sequential boost (15 x 2.67 Gy WBI + 6 x 2.48 Gy boost)
  Arms: Minimal surgical margin <1 mm, conventional arm: seq boost
Radiation: SIB (15 x 2.67 Gy WBI and SIB 15 x 2.67-3.33 Gy) — Minimal surgical margin < 1 mm, experimental arm with SIB (15 x 2.67 Gy WBI and SIB 15 x 2.67-3.33 Gy)
  Arms: Minimal surgical margin < 1 mm, experimental arm with SIB.

SUMMARY:
Whole breast irradiation (WBI) after breast conserving surgery for early-stage breast cancer halves the recurrence risk and reduces the breast cancer death by about one sixth. A sequential boost (SeqB) dose to the tumour bed further improves local control, but also increases the risk of late skin toxicity and cosmetic changes. At Ghent University Hospital WBI is prescribed in 15 fractions of 2.67 Gy according to the START-B hypofractionation scheme. A sequential boost is typically given in 4 to 8 extra fractions which prolongs the overall treatment time. The boost dose can also be delivered within the 15 fractions of WBI, the so-called simultaneous integrated boost (SIB). SIB shortens the overall treatment time which is convenient for the patient and the radiotherapy department. In this study we wish to test the hypothesis of acceptable skin toxicity and reduced cost with SIB using hypofractionated prone intensity modulation radiotherapy IMRT with topographical dose painting, a technique recently developed in our group. Patients are randomized between SeqB and SIB.

ELIGIBILITY:
Inclusion criteria:

Female patients AND breast conserving surgery AND multidisciplinary decision of adjuvant WBI with a boost to the tumor bed AND age ≥ 18 years AND informed consent obtained, signed and dated before specific protocol procedures

Exclusion criteria

* Mastectomy
* Need for lymph node irradiation
* No boost
* Bilateral breast irradiation
* Patient not able to reach or maintain the prone position
* Pregnant or breastfeeding
* Mental condition rendering the patient unable to understand the nature, scope and possible consequences of the study
* Patient unlikely to comply with the protocol; i.e. uncooperative attitude, inability to return for follow-up visits, and unlikely to complete the study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2012-12 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2021-03 (Actual)

PRIMARY OUTCOMES:
Degree of acute moist desquamation during or in the first 2 weeks after radiotherapy. | weekly during radiotherapy, 2 weeks after the end of radiotherapy.
  Clinical inspection of the treated breast.

SECONDARY OUTCOMES:
Degree of acute skin toxicity. | Weekly during radiotherapy and 2 weeks after the end of radiotherapy.
  Clinical inspection.
Degree of chronic skin toxicity and cosmesis after radiotherapy. | 2 weeks, 1 year, 2 years and 5 years after radiotherapy.
  Inspection, clinical evaluation, digital photographs.
Quality of life after radiotherapy. | 2 weeks, 1 year, 2 years and 5 years after radiotherapy.
  QLQ C30 and QLQ BR23 quality of life questionnaires.
Biomarker analysis. | Blood sample within 1 week before the start of radiotherapy
  Blood sample
Measurement of costs for the patient for the full treatment. | Over the period of radiotherapy treatment, with a maximum of 5 weeks.
  Activity based costing models.

CONTACTS AND LOCATIONS:
Overall Officials: Wilfried De Neve, MD, PhD, Principal Investigator — University Hospital, Ghent
Locations (1):
- Ghent University Hospital, Ghent, Belgium

REFERENCES:
- See also: Related Info — http://www.uzgent.be